CLINICAL TRIAL: NCT01307267
Title: A PHASE 1 STUDY OF PF-05082566 AS A SINGLE AGENT IN PATIENTS WITH ADVANCED CANCER, AND IN COMBINATION WITH RITUXIMAB IN PATIENTS WITH NON-HODGKIN'S LYMPHOMA (NHL)
Brief Title: A Study Of PF-05082566 As A Single Agent And In Combination With Rituximab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1641001; 2011-002799-17 (EudraCT Number)
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Carcinoma, Squamous Cell of Head and Neck; Malignant Melanoma
Keywords: Phase 1; Non-Hodgkin's Lymphoma; Advanced malignancies
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Squamous Cell Carcinoma of Head and Neck; Melanoma | interventions — utomilumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Portion A (Experimental): PF-05082566 single agent in patients with advanced cancer
  Interventions: Drug: PF-05082566
- Portion B (Experimental): PF-05082566 in combination with rituximab in patients with Non-Hodgkin's Lymphoma
  Interventions: Drug: rituximab; Drug: PF-05082566

INTERVENTIONS:
Drug: PF-05082566 — Intravenous, Dose escalation, once per month
  Arms: Portion A
Drug: rituximab — Intravenous, 375 mg/m2, once per week for 4 weeks
  Other Names: Rituxan, MabThera
  Arms: Portion B
Drug: PF-05082566 — IV, Dose escalation, once per month
  Arms: Portion B

SUMMARY:
A study of PF-05082566, a 4-1BB agonist monoclonal antibody (mAb), in patients with solid tumors or b-cell lymphomas, and in combination with rituximab in patients with CD20 positive Non-Hodgkin's Lymphoma (NHL).

ELIGIBILITY:
Inclusion Criteria

* Portion A: Histological or cytological diagnosis of advanced/metastatic solid tumor malignancy or B cell lymphoma, for which no curative therapy is available. Portion A expansion includes patients who have documented disease progression on a checkpoint inhibitor (anti CTLA 4, anti PD1/PD L1 antibodies) per RECIST criteria. Tumor types include metastatic melanoma, renal cell carcinoma (RCC), non-small cell lung cancer (NCSLC) and squamous cell carcinoma of the head and neck (SCCHN). Patients in the dose expansion stage are required to provide archival or baseline (obtained during the screening period) tumor biopsies.
* Portion B: Histological confirmed relapsed or refractory CD20 positive NHL for which no curative therapy is available. Patients enrolled in the expansion cohort must have archival tissue available, sampled within 6 months of study entry. The Expansion cohort includes patients with FL or DLBCL with relapsed or refractory disease.
* Measurable disease with at least one extranodal tumor mass >1.0 cm in the greatest transverse diameter (GTD) or in the case of malignant lymph nodes >1.5 cm in the GTD.
* ECOG performance status of ≤ 1.
* Adequate bone marrow function, for Portion A: absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥100 x 109/L, hemoglobin >9.0 g/dL. For Portion B: ANC ≥ 1.0 x 109/L, platelet count ≥ 75 x 109/L, and hemoglobin ≥ 8.0 g/dL. In both cases, patients must be transfusion independent at least 14 days prior to screening.
* Serum creatinine ≤ 2 x ULN or estimated creatinine clearance ≥ 50 ml/min.
* Total serum bilirubin ≤ 1.5 x ULN unless the patient has documented Gilbert syndrome and AST and ALT ≤ 2.5 x ULN.

Exclusion Criteria

* Patients with known symptomatic brain metastases requiring steroids.
* Prior allogeneic hematopoietic stem cell transplant.
* Immunosuppressive regimens involving systemic corticosteroids within 14 days before the first dose of study treatment.
* Therapeutic or experimental monoclonal antibodies within 28 day or prior radiation therapy within 14 days of the first dose of study drug.
* Autoimmune disorders and other diseases that compromise or impair the immune system.
* Unstable or serious concurrent medical conditions in the previous 6 months.
* Prior therapy with any anti CD137 monoclonal antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2011-06-21 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- United States (33):
  - City of Hope, Duarte, California
  - UC San Diego Moores Cancer Center-Investigational Drug Services, La Jolla, California
  - UC San Diego Medical Center-La Jolla (Jacobs Medical Center/Thornton Hospital), La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Research Administration Office: Clinical Research Unit, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Drug Information Center, Los Angeles, California
  - UCLA Bowyer Clinic, Los Angeles, California
  - UCLA Hematology-Oncology Clinic, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Santa Monica UCLA Hematology & Oncology Clinic, Santa Monica, California
  - Stanford University Medical Center, Stanford, California
  - Georgetown University Medical Center Department of Pharmacy, Research, Washington D.C., District of Columbia
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - The Emory Clinic, Building A, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Brigham and Woman's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Siteman Cancer Center - St. Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center-West County, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University Infusion Center Pharmacy, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center- South County, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The University of Texas - M.D. Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- Centre d'investigation clinique, Rennes, France
- Italy (2):
  - Az. Ospedaliera-Univer. di Bologna Policlinico S. Orsola Malpighi, Bologna, BO
  - Ospedale San Raffaele di Milano, Milan, MI
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Akita University Hospital, Akita
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Tokyo

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Gopal AK, Levy R, Houot R, Patel SP, Popplewell L, Jacobson C, Mu XJ, Deng S, Ching KA, Chen Y, Davis CB, Huang B, Fly KD, Thall A, Woolfson A, Bartlett NL. First-in-Human Study of Utomilumab, a 4-1BB/CD137 Agonist, in Combination with Rituximab in Patients with Follicular and Other CD20+ Non-Hodgkin Lymphomas. Clin Cancer Res. 2020 Jun 1;26(11):2524-2534. doi: 10.1158/1078-0432.CCR-19-2973. Epub 2020 Mar 6. PMID 32144134
- [Derived] Segal NH, He AR, Doi T, Levy R, Bhatia S, Pishvaian MJ, Cesari R, Chen Y, Davis CB, Huang B, Thall AD, Gopal AK. Phase I Study of Single-Agent Utomilumab (PF-05082566), a 4-1BB/CD137 Agonist, in Patients with Advanced Cancer. Clin Cancer Res. 2018 Apr 15;24(8):1816-1823. doi: 10.1158/1078-0432.CCR-17-1922. Epub 2018 Mar 16. PMID 29549159
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1641001&StudyName=A%20Study%20Of%20PF-05082566%20As%20A%20Single%20Agent%20And%20In%20Combination%20With%20Rituximab

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was 1 participant who was enrolled but withdrew the consent before starting any of the treatment arms; therefore, this participant was not included in the participant flow table.
Groups:
- Portion A: PF-05082566 0.006mg/kg: Participants received PF-05082566 0.006 milligrams per kilogram (mg/kg) intravenously once every 4 weeks (q4wks) as a single agent in Portion A, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion A: PF-05082566 0.03mg/kg: Participants received PF-05082566 0.03mg/kg intravenously q4wks as a single agent in Portion A, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion A: PF-05082566 0.06mg/kg: Participants received PF-05082566 0.06mg/kg intravenously q4wks as a single agent in Portion A, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion A: PF-05082566 0.12mg/kg: Participants received PF-05082566 0.12mg/kg intravenously q4wks as a single agent in Portion A, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion A: PF-05082566 0.18mg/kg: Participants received PF-05082566 0.18mg/kg intravenously q4wks as a single agent in Portion A, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion A: PF-05082566 0.24mg/kg: Participants received PF-05082566 0.24mg/kg intravenously q4wks as a single agent in Portion A, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion A: PF-05082566 0.3mg/kg: Participants received PF-05082566 0.3mg/kg intravenously q4wks as a single agent in Portion A, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion A: PF-05082566 0.6mg/kg: Participants received PF-05082566 0.6mg/kg intravenously q4wks as a single agent in Portion A, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion A: PF-05082566 1.2mg/kg: Participants received PF-05082566 1.2mg/kg intravenously q4wks as a single agent in Portion A, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion A: PF-05082566 2.4mg/kg: Participants received PF-05082566 2.4mg/kg intravenously q4wks as a single agent in Portion A, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion A: PF-05082566 5mg/kg: Participants received PF-05082566 5mg/kg intravenously q4wks as a single agent in Portion A, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion A: PF-05082566 10mg/kg: Participants received PF-05082566 10mg/kg intravenously q4wks as a single agent in Portion A, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2: Participants received PF-05082566 0.03mg/kg intravenously q4wks in combination with rituximab (375 milligrams per square meter [mg/m^2] intravenously, every week during the first 4 weeks) in Portion B, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2: Participants received PF-05082566 0.06mg/kg intravenously q4wks in combination with rituximab (375mg/m^2 intravenously, every week during the first 4 weeks) in Portion B, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2: Participants received PF-05082566 0.12mg/kg intravenously q4wks in combination with rituximab (375mg/m^2 intravenously, every week during the first 4 weeks) in Portion B, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2: Participants received PF-05082566 0.18mg/kg intravenously q4wks in combination with rituximab (375mg/m^2 intravenously, every week during the first 4 weeks) in Portion B, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2: Participants received PF-05082566 0.24mg/kg intravenously q4wks in combination with rituximab (375mg/m^2 intravenously, every week during the first 4 weeks) in Portion B, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2: Participants received PF-05082566 0.3mg/kg intravenously q4wks in combination with rituximab (375mg/m^2 intravenously, every week during the first 4 weeks) in Portion B, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2: Participants received PF-05082566 0.6mg/kg intravenously q4wks in combination with rituximab (375mg/m^2 intravenously, every week during the first 4 weeks) in Portion B, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2: Participants received PF-05082566 1.2mg/kg intravenously q4wks in combination with rituximab (375mg/m^2 intravenously, every week during the first 4 weeks) in Portion B, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2: Participants received PF-05082566 2.4mg/kg intravenously q4wks in combination with rituximab (375mg/m^2 intravenously, every week during the first 4 weeks) in Portion B, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2: Participants received PF-05082566 5mg/kg intravenously q4wks in combination with rituximab (375mg/m^2 intravenously, every week during the first 4 weeks) in Portion B, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
- Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2: Participants received PF-05082566 10mg/kg intravenously q4wks in combination with rituximab (375mg/m^2 intravenously, every week during the first 4 weeks) in Portion B, for up to 2 years or until participant permanently discontinued study treatment, whichever occurred earlier.
Period: Overall Study
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Started | 4 | 3 | 6 | 4 | 3 | 42 | 3 | 4 | 31 | 5 | 6 | 11 | 3 | 3 | 4 | 3 | 3 | 3 | 4 | 32 | 3 | 5 | 4
Completed | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 5 | 3 | 1 | 41 | 2 | 4 | 30 | 5 | 6 | 11 | 1 | 0 | 2 | 1 | 1 | 1 | 2 | 32 | 3 | 5 | 4
Not completed — Death | 4 | 3 | 5 | 3 | 1 | 26 | 2 | 2 | 21 | 2 | 3 | 9 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 8 | 1 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 5 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 1 | 3 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 19 | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of PF-05082566 or rituximab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2 | Total
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 42 | 3 | 4 | 31 | 5 | 6 | 11 | 3 | 3 | 4 | 3 | 3 | 3 | 4 | 32 | 3 | 5 | 4 | 189
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 4 | 3 | 1 | 17 | 1 | 2 | 19 | 4 | 3 | 5 | 3 | 2 | 4 | 0 | 2 | 3 | 2 | 14 | 0 | 3 | 3 | 100
  >=65 years | 1 | 1 | 2 | 1 | 2 | 25 | 2 | 2 | 12 | 1 | 3 | 6 | 0 | 1 | 0 | 3 | 1 | 0 | 2 | 18 | 3 | 2 | 1 | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 2 | 2 | 15 | 0 | 1 | 13 | 3 | 1 | 3 | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 15 | 1 | 2 | 1 | 72
  Male | 4 | 2 | 4 | 2 | 1 | 27 | 3 | 3 | 18 | 2 | 5 | 8 | 1 | 2 | 2 | 2 | 1 | 2 | 3 | 17 | 2 | 3 | 3 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 3 | 4 | 2 | 36 | 1 | 4 | 24 | 4 | 2 | 4 | 2 | 3 | 3 | 2 | 2 | 2 | 4 | 22 | 2 | 5 | 4 | 141
  Black | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 7
  Asian | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 22
  Other | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 4 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 18
  Unspecified | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs) in First 2 Cycles of Portion A
Description: DLT: Any of the following adverse events (AEs) occurred in the first 2 cycles of treatment (up to 28 days post second dose) which was attributed to PF-05082566 alone for Portion A and not related to progressive disease. Hematologic: Grade 4 neutropenia lasting more than (>)7 days; febrile neutropenia; neutropenic infection; Grade ≥3 thrombocytopenia with bleeding; Grade 4 thrombocytopenia; Grade ≥3 hemolysis. Non-Hematologic: Grade ≥3 toxicities, except those Grade 3 events that responded to treatment (eg, Grade 3 nausea, vomiting, diarrhea responding to standard medical supportive care within 48 hours would not be considered a DLT). Severity of AEs were graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 (Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death related to AE). Each cycle=28 days.
Time Frame: Cycle 1 Day 1 to Cycle 2 Day 29 in Portion A (up to 57 days, each cycle = 28 days)
Population: All participants who received at least 1 dose of PF-05082566 in the first 2 cycles of Portion A.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 42 | 3 | 4 | 31 | 5 | 6 | 11
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With DLTs in First 2 Cycles of Portion B
Description: DLT: Any of the following AEs occurred in the first 2 cycles of treatment (up to 28 days post second dose) which was attributed to PF-05082566 in combination with rituximab for Portion B and not related to progressive disease. Hematologic: Grade 4 neutropenia lasting more than (>)7 days; febrile neutropenia; neutropenic infection; Grade ≥3 thrombocytopenia with bleeding; Grade 4 thrombocytopenia; Grade ≥3 hemolysis. Non-Hematologic: Grade ≥3 toxicities, except those Grade 3 events that responded to treatment (eg, Grade 3 nausea, vomiting, diarrhea responding to standard medical supportive care within 48 hours would not be considered a DLT). Severity of AEs were graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 (Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death related to AE). Each cycle=28 days.
Time Frame: Cycle 1 Day 1 to Cycle 2 Day 29 in Portion B (up to 57 days, each cycle = 28 days)
Population: All participants who received at least 1 dose of PF-05082566 and 1 dose of rituximab in the first 2 cycles of Portion B.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 31 | 3 | 5 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) in Portion A
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. AEs included both non-serious AEs and SAEs. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study treatment. Causality of AEs was determined by the investigator.
Time Frame: Up to approximately 2 years
Population: All participants who received at least 1 dose of PF-05082566 in Portion A.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 42 | 3 | 4 | 31 | 5 | 6 | 11
Participants
  AEs | 3 | 3 | 5 | 4 | 3 | 39 | 3 | 4 | 26 | 5 | 5 | 9
  SAEs | 0 | 0 | 2 | 1 | 0 | 13 | 0 | 0 | 8 | 1 | 2 | 3
  AEs related to PF-05082566 | 2 | 1 | 2 | 1 | 2 | 25 | 1 | 1 | 10 | 1 | 2 | 4
  SAEs related to PF-05082566 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Treatment-Emergent AEs by Maximum National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE) Grade in Portion A
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study treatment. Severity of AEs were graded according to NCI CTCAE version 4.03 (Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death related to AE).
Time Frame: Up to approximately 2 years
Population: All participants who received at least 1 dose of PF-05082566 in Portion A.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 42 | 3 | 4 | 31 | 5 | 6 | 11
Participants
  Grade 1 | 0 | 0 | 1 | 1 | 1 | 9 | 2 | 1 | 7 | 1 | 1 | 2
  Grade 2 | 1 | 2 | 2 | 1 | 0 | 14 | 1 | 2 | 8 | 3 | 2 | 4
  Grade 3 | 2 | 1 | 2 | 2 | 2 | 12 | 0 | 1 | 9 | 1 | 2 | 2
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1

5. Secondary Outcome: Number of Participants With Hematology Laboratory Abnormalities by Maximum NCI CTCAE Grade in Portion A
Description: Following hematology laboratory abnormalities were graded per NCI CTCAE version 4.03: anemia, hemoglobin increased, lymphocyte count increased, lymphopenia, neutrophils (absolute), platelets, white blood cells. The abnormalities with at least 1 participant are presented here.
Time Frame: Up to approximately 2 years
Population: All participants who received at least 1 dose of PF-05082566 in Portion A and had hematology laboratory test data.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 42 | 3 | 4 | 28 | 4 | 6 | 11
Participants
  Anemia, Grade 1 | 1 | 3 | 3 | 3 | 1 | 20 | 2 | 1 | 12 | 1 | 3 | 6
  Anemia, Grade 2 | 2 | 0 | 3 | 1 | 1 | 6 | 0 | 2 | 8 | 0 | 2 | 5
  Anemia, Grade 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Lymphocyte count increased, Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphopenia, Grade 1 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 1 | 4 | 1 | 0 | 6
  Lymphopenia, Grade 2 | 3 | 0 | 2 | 0 | 2 | 10 | 1 | 1 | 6 | 1 | 3 | 2
  Lymphopenia, Grade 3 | 1 | 1 | 1 | 3 | 1 | 7 | 1 | 1 | 2 | 1 | 1 | 0
  Lymphopenia, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (absolute), Grade 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
  Neutrophils (absolute), Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Neutrophils (absolute), Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Platelets, Grade 1 | 2 | 2 | 2 | 1 | 2 | 7 | 1 | 2 | 2 | 1 | 1 | 1
  White blood cells, Grade 1 | 1 | 1 | 1 | 2 | 0 | 4 | 1 | 2 | 6 | 0 | 2 | 3
  White blood cells, Grade 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White blood cells, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Chemistries Laboratory Abnormalities by Maximum NCI CTCAE Grade in Portion A
Description: Following chemistries laboratory abnormalities were graded per NCI CTCAE version 4.03: alanine aminotransferase (ALT), Alkaline phosphatase, Aspartate aminotransferase (AST), bilirubin (total), creatinine, gamma glutamyl transferase (GGT), hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, hypophosphatemia. The abnormalities with at least 1 participant are presented here.
Time Frame: Up to approximately 2 years
Population: "Number of Participants Analyzed" represents all participants who received at least 1 dose of PF-05082566 in Portion A and had chemistries laboratory test data. "Number Analyzed" represents all participants who received at least 1 dose of PF-05082566 in Portion A and had data for the specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 42 | 3 | 4 | 28 | 4 | 6 | 11
Participants
  ALT, Grade 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 6 | 0 | 0 | 1
  ALT, Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Alkaline phosphatase, Grade 1 | 2 | 0 | 1 | 0 | 2 | 13 | 0 | 0 | 6 | 1 | 3 | 4
  Alkaline phosphatase, Grade 2 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 2 | 0 | 0 | 0
  Alkaline phosphatase, Grade 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Grade 1 | 3 | 2 | 1 | 1 | 2 | 12 | 2 | 2 | 7 | 1 | 2 | 1
  AST, Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin (total), Grade 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
  Bilirubin (total), Grade 2 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine, Grade 1 | 3 | 3 | 5 | 4 | 3 | 22 | 2 | 2 | 19 | 4 | 5 | 6
  Creatinine, Grade 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1
  GGT, Grade 2: number analyzed (Participants) | 4 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GGT, Grade 2 | 1 | 0 | 1 |  |  |  |  |  |  |  |  |
  GGT, Grade 3: number analyzed (Participants) | 4 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GGT, Grade 3 | 1 | 2 | 1 |  |  |  |  |  |  |  |  |
  Hypercalcemia, Grade 1 | 1 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 1 | 0 | 0
  Hyperglycemia, Grade 1 | 2 | 0 | 3 | 3 | 3 | 20 | 3 | 3 | 13 | 2 | 4 | 6
  Hyperglycemia, Grade 2 | 2 | 2 | 2 | 0 | 0 | 7 | 0 | 1 | 3 | 1 | 1 | 3
  Hyperglycemia, Grade 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
  Hyperkalemia, Grade 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 3 | 1 | 0 | 0
  Hyperkalemia, Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia, Grade 1: number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 42 | 3 | 4 | 27 | 4 | 6 | 11
  Hypermagnesemia, Grade 1 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 3 | 0 | 1 | 0
  Hypermagnesemia, Grade 3: number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 42 | 3 | 4 | 27 | 4 | 6 | 11
  Hypermagnesemia, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypernatremia, Grade 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Hypoalbuminemia, Grade 1 | 1 | 1 | 4 | 4 | 1 | 18 | 1 | 3 | 9 | 2 | 2 | 4
  Hypoalbuminemia, Grade 2 | 2 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 1 | 4
  Hypoalbuminemia, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia, Grade 1 | 1 | 0 | 0 | 0 | 0 | 7 | 0 | 1 | 5 | 0 | 3 | 0
  Hypocalcemia, Grade 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypoglycemia, Grade 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Hypoglycemia, Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypokalemia, Grade 1 | 1 | 0 | 2 | 1 | 1 | 4 | 2 | 1 | 3 | 1 | 0 | 2
  Hypokalemia, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Hypokalemia, Grade 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia, Grade 1: number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 42 | 3 | 4 | 27 | 4 | 6 | 11
  Hypomagnesemia, Grade 1 | 2 | 1 | 1 | 2 | 0 | 8 | 0 | 1 | 3 | 1 | 1 | 0
  Hyponatremia, Grade 1 | 2 | 2 | 2 | 1 | 0 | 17 | 2 | 0 | 8 | 4 | 1 | 2
  Hyponatremia, Grade 3 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0
  Hypophosphatemia, Grade 2: number analyzed (Participants) | 4 | 3 | 5 | 3 | 3 | 40 | 3 | 4 | 27 | 4 | 6 | 11
  Hypophosphatemia, Grade 2 | 0 | 2 | 0 | 2 | 0 | 8 | 2 | 0 | 0 | 0 | 0 | 3
  Hypophosphatemia, Grade 3: number analyzed (Participants) | 4 | 3 | 5 | 3 | 3 | 40 | 3 | 4 | 27 | 4 | 6 | 11
  Hypophosphatemia, Grade 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Vital Sign Abnormalities in Portion A
Description: For vital signs in Portion A, blood pressure and pulse rate were measured. Clinical significance was determined by the investigator.
Time Frame: Up to approximately 2 years
Population: All participants who received at least 1 dose of PF-05082566 in Portion A.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 42 | 3 | 4 | 31 | 5 | 6 | 11
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: PF-05082566 Maximum Observed Serum Concentration (Cmax) in Portion A
Description: Cmax of PF-05082566 was observed directly from data.
Time Frame: Day 1 of Cycle 1 and Cycle 2 at pre-dose, and 1, 1.5, 2, 6, 24, 48, 168, 336 and 504 hours post-dose
Population: All participants who received at least 1 dose of PF-05082566 in Portion A and had at least 1 of the PK parameters of interest. "Number Analyzed" represents those participants who had data for each specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 40 | 3 | 4 | 29 | 5 | 6 | 11
micrograms per milliliter (μg/mL)
  Cycle 1 | 0.1515 (12) | 0.4952 (34) | 1.014 (24) | 2.614 (23) | 4.219 (16) | 3.246 (30) | 7.038 (23) | 11.72 (28) | 18.02 (24) | 49.63 (24) | 97.75 (13) | 150.3 (24)
  Cycle 2: number analyzed (Participants) | 2 | 3 | 6 | 3 | 3 | 37 | 2 | 4 | 24 | 3 | 5 | 10
  Cycle 2 | 0.1250 (NA) — Geometric coefficient of variation (CV) was not calculated when there were less than 3 participants with data. | 0.5049 (7) | 1.093 (47) | 3.408 (25) | 4.013 (25) | 2.955 (46) | 8.349 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 14.80 (24) | 17.61 (36) | 58.38 (33) | 101.6 (17) | 167.0 (21)

9. Secondary Outcome: PF-05082566 Pre-dose Trough Concentration During Multiple Dosing (Ctrough) in Portion A
Description: Ctrough of PF-05082566 was observed directly from data.
Time Frame: Day 1 pre-dose of Cycle 2
Population: All participants who received at least 1 dose of PF-05082566 in Portion A and had data for Ctrough.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 2 | 3 | 6 | 3 | 3 | 37 | 2 | 4 | 24 | 3 | 5 | 10
μg/mL | NA (NA) — Geometric mean cannot be calculated when there were participants with a zero value (ie, Ctrough below the limit of quantification). Geometric CV was not calculated when there were less than 3 participants with data. | 0.1063 (24) | 0.1092 (24) | 0.3268 (12) | 0.4285 (49) | 0.3868 (46) | 0.8597 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 1.520 (22) | 1.313 (61) | 7.054 (52) | 9.934 (35) | 9.963 (250)

10. Secondary Outcome: PF-05082566 Time for Maximum Observed Serum Concentration (Tmax) in Portion A
Description: Tmax of PF-05082566 was observed directly from data as time of Cmax.
Time Frame: Day 1 of Cycle 1 and Cycle 2 at pre-dose, and 1, 1.5, 2, 6, 24, 48, 168, 336 and 504 hours post-dose.
Population: as for outcome 8
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 40 | 3 | 4 | 29 | 5 | 6 | 11
hours (hr)
  Cycle 1 | 1.75 [1.50 to 2.00] | 1.63 [1.50 to 1.67] | 2.00 [1.00 to 5.42] | 1.26 [1.00 to 2.00] | 1.25 [0.967 to 6.00] | 1.03 [0.833 to 24.2] | 1.00 [1.00 to 1.50] | 1.80 [1.62 to 2.00] | 1.17 [1.00 to 5.53] | 1.50 [1.00 to 1.58] | 1.06 [1.00 to 1.48] | 1.50 [1.07 to 2.02]
  Cycle 2: number analyzed (Participants) | 2 | 3 | 6 | 3 | 3 | 37 | 2 | 4 | 24 | 3 | 5 | 10
  Cycle 2 | 13.0 [2.00 to 24.0] | 1.50 [1.50 to 2.00] | 1.54 [1.00 to 2.00] | 1.00 [1.00 to 2.00] | 2.00 [1.50 to 2.00] | 1.03 [0.833 to 2.00] | 1.00 [1.00 to 1.00] | 1.46 [1.00 to 1.70] | 1.02 [0.883 to 1.22] | 1.08 [1.00 to 1.08] | 1.92 [1.08 to 2.00] | 1.31 [1.03 to 5.55]

11. Secondary Outcome: PF-05082566 Area Under the Serum Concentration-Time Profile (AUC) From Time 0 to the Time of the Last Measurable Concentration (AUClast) in Portion A
Description: AUClast of PF-05082566 was determined by linear/log trapezoidal method.
Time Frame: Day 1 of Cycle 1 and Cycle 2 at pre-dose, and 1, 1.5, 2, 6, 24, 48, 168, 336 and 504 hours post-dose.
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (μg*hr/mL)
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 40 | 3 | 4 | 29 | 5 | 6 | 11
microgram*hour per milliliter (μg*hr/mL)
  Cycle 1: number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 34 | 3 | 4 | 27 | 5 | 6 | 11
  Cycle 1 | 8.212 (251) | 101.0 (9) | 148.1 (33) | 389.4 (58) | 703.3 (32) | 481.1 (48) | 996.1 (29) | 2165 (21) | 2383 (61) | 5731 (101) | 15540 (22) | 25520 (24)
  Cycle 2: number analyzed (Participants) | 2 | 3 | 6 | 3 | 3 | 5 | 2 | 4 | 4 | 3 | 5 | 10
  Cycle 2 | 14.21 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 105.2 (49) | 93.59 (152) | 614.9 (7) | 808.0 (53) | 818.7 (38) | 1662 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 1918 (40) | 4035 (25) | 6741 (6) | 18140 (24) | 19900 (51)

12. Secondary Outcome: PF-05082566 AUC From Time 0 to Infinity (AUCinf) in Portion A
Description: AUCinf = AUClast + (Clast*/kel), where Clast* is the estimated concentration at the time of the last measurable concentration and kel is the terminal phase rate constant calculated as the absolute value of the slope of a linear regression during the terminal phase of the natural log-transformed concentration time profile.
Time Frame: Day 1 of Cycle 1 and Cycle 2 at pre-dose, and 1, 1.5, 2, 6, 24, 48, 168, 336 and 504 hours post-dose.
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 40 | 3 | 4 | 29 | 5 | 6 | 11
μg*hr/mL
  Cycle 1: number analyzed (Participants) | 0 | 1 | 6 | 3 | 2 | 15 | 1 | 2 | 21 | 2 | 4 | 8
  Cycle 1 |  | 120 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 187.5 (31) | 667.0 (13) | 989.5 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 687.9 (43) | 770.0 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 2916 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 3111 (36) | 7628 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 18430 (24) | 28280 (28)
  Cycle 2: number analyzed (Participants) | 0 | 2 | 3 | 1 | 3 | 5 | 1 | 2 | 3 | 1 | 3 | 3
  Cycle 2 |  | 169.8 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 251.4 (17) | 931.0 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 1072 (57) | 960.8 (47) | 2000 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 1782 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 4649 (25) | 8480 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 20950 (23) | 22400 (26)

13. Secondary Outcome: PF-05082566 AUC From Time 0 to Time of Dosing Interval (AUCtau) in Portion A
Description: AUCtau of PF-05082566 was determined using linear/log trapezoidal method.
Time Frame: Day 1 of Cycle 1 and Cycle 2 at pre-dose, and 1, 1.5, 2, 6, 24, 48, 168, 336 and 504 hours post-dose.
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 40 | 3 | 4 | 29 | 5 | 6 | 11
μg*hr/mL
  Cycle 1: number analyzed (Participants) | 4 | 3 | 6 | 3 | 3 | 32 | 3 | 4 | 25 | 4 | 6 | 11
  Cycle 1 | 13.70 (181) | 104.8 (9) | 154.2 (27) | 503.9 (14) | 690.9 (33) | 538.6 (33) | 1012 (27) | 2195 (21) | 2761 (34) | 8204 (36) | 15760 (20) | 25250 (23)
  Cycle 2: number analyzed (Participants) | 0 | 2 | 3 | 2 | 3 | 5 | 2 | 3 | 4 | 1 | 5 | 4
  Cycle 2 |  | 130.8 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 224.4 (19) | 618.6 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 864.1 (47) | 824.3 (37) | 1681 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 2107 (43) | 4068 (27) | 7460 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 19040 (18) | 20490 (17)

14. Secondary Outcome: PF-05082566 Clearance (CL) in Portion A
Description: CL = Dose/AUCinf for Cycle 1 and Dose/AUCtau for Cycle 2. It was reported in units of milliliter per hour per kilogram (mL/hr/kg).
Time Frame: Day 1 of Cycle 1 and Cycle 2 at pre-dose, and 1, 1.5, 2, 6, 24, 48, 168, 336 and 504 hours post-dose.
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/hour/kilogram (mL/hr/kg)
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 40 | 3 | 4 | 29 | 5 | 6 | 11
milliliter/hour/kilogram (mL/hr/kg)
  Cycle 1: number analyzed (Participants) | 0 | 1 | 6 | 3 | 2 | 15 | 1 | 2 | 21 | 2 | 4 | 8
  Cycle 1 |  | 0.2510 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.3203 (31) | 0.1800 (13) | 0.1823 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.3490 (42) | 0.3890 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.2054 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.3861 (36) | 0.3145 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.2711 (24) | 0.3536 (28)
  Cycle 2: number analyzed (Participants) | 0 | 2 | 3 | 2 | 3 | 5 | 2 | 3 | 4 | 1 | 5 | 4
  Cycle 2 |  | 0.2296 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.2676 (19) | 0.1939 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.2082 (47) | 0.2906 (37) | 0.1786 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.2847 (43) | 0.2950 (27) | 0.3220 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.2626 (18) | 0.4883 (17)

15. Secondary Outcome: PF-05082566 Volume of Distribution at Steady State (Vss) in Portion A
Description: Vss = CL × MRT, where CL is clearance and MRT is the mean residence time after intravenous administration.
Time Frame: Day 1 of Cycle 1 and Cycle 2 at pre-dose, and 1, 1.5, 2, 6, 24, 48, 168, 336 and 504 hours post-dose.
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per kilogram (mL/kg)
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 40 | 3 | 4 | 29 | 5 | 6 | 11
milliliter per kilogram (mL/kg)
  Cycle 1: number analyzed (Participants) | 0 | 1 | 6 | 3 | 2 | 15 | 1 | 2 | 21 | 2 | 4 | 8
  Cycle 1 |  | 65.50 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 101.1 (20) | 83.63 (15) | 74.38 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 110.7 (28) | 75.20 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 82.38 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 112.2 (29) | 110.4 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 97.07 (26) | 125.5 (21)
  Cycle 2: number analyzed (Participants) | 0 | 2 | 3 | 1 | 3 | 5 | 1 | 2 | 3 | 1 | 3 | 3
  Cycle 2 |  | 102.1 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 74.11 (21) | 90.80 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 81.69 (27) | 86.50 (29) | 51.00 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 61.54 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 116.5 (62) | 99.80 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 87.37 (43) | 139.5 (29)

16. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) for PF-05082566 in Portion A
Description: ADA for PF-05082566 was detected using electrochemiluminescence assay. Positive ADA for PF-05082566: titer>=6.23.
Time Frame: Up to approximately 2 years
Population: All participants who received at least 1 dose of PF-05082566 in Portion A and was tested for ADA.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 42 | 3 | 4 | 31 | 5 | 6 | 11
Participants | 4 | 2 | 5 | 0 | 0 | 20 | 1 | 3 | 14 | 1 | 3 | 2

17. Secondary Outcome: Number of Participants With QTc Interval Meeting Categorical Summarization Criteria in Portion A
Description: Categorical summarization criteria for QTc interval (time from ECG Q wave to the end of the T wave corresponding to electrical systole corrected for heart rate): 1) absolute value of >450 to <=480 milliseconds (msec), >480 to <=500 msec, >500 msec; 2) a maximum change from baseline of >30 to <=60 msec or >60 msec.
Time Frame: Up to approximately 2 years
Population: All participants who received at least 1 dose of PF-05082566 in Portion A and had post-baseline QTc data. "Number Analyzed" represents those participants who had data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 40 | 3 | 4 | 29 | 5 | 6 | 11
Participants
  QTc >450 to <=480 msec | 1 | 0 | 0 | 2 | 0 | 10 | 0 | 1 | 8 | 2 | 3 | 4
  QTc >480 to <=500 msec | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
  QTc >500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  QTc change >30 to <=60 msec: number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 39 | 3 | 4 | 29 | 5 | 6 | 11
  QTc change >30 to <=60 msec | 0 | 0 | 0 | 0 | 1 | 6 | 0 | 0 | 0 | 0 | 2 | 3
  QTc change >60 msec: number analyzed (Participants) | 4 | 3 | 6 | 4 | 3 | 39 | 3 | 4 | 29 | 5 | 6 | 11
  QTc change >60 msec | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Percentage of Participants Achieving Objective Response Per Response Evaluation Criteria in Solid Tumor (RECIST) Version 1.1 in Portion A
Description: Objective response: confirmed best overall response (BOR) of complete response (CR) or partial response (PR) per RECIST version 1.1. BOR of CR: target lesions and non-target diseases achieved CR, without new lesions. BOR of PR: target lesions achieved CR or PR while non-target diseases were non-CR/non-progression of disease (non-PD), indeterminate or missing, and without new lesions. For target lesions, CR: complete disappearance of all target lesions except nodal disease (target nodes must decrease to normal size); PR: >=30% decrease under baseline of the sum of diameters of all target measurable lesions. For non-target diseases, CR: disappearance of all non-target lesions and normalization of tumor marker levels; non-CR/non-PD: persistence of any non-target lesions and/or tumor marker level above the normal limits; Indeterminate: progression had not been determined and >=1 non-target sites were not assessed or assessment methods were inconsistent with those used at baseline.
Time Frame: Every 8 weeks from Cycle 1 Day 1 for the first 10 months on study treatment, then every 16 weeks till follow-up visit (assessed up to approximately 2 years)
Population: All participants who received at least 1 dose of PF-05082566 in Portion A and had tumor assessments.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 1 | 42 | 3 | 4 | 31 | 5 | 6 | 11
percentage of participants | 0 [0 to 60.2] | 0 [0 to 70.8] | 0 [0 to 45.9] | 0 [0 to 60.2] | 0 [0 to 97.5] | 4.8 [0.6 to 16.2] | 0 [0 to 70.8] | 25.0 [0.6 to 80.6] | 0 [0 to 11.2] | 0 [0 to 52.2] | 0 [0 to 45.9] | 0 [0 to 28.5]

19. Secondary Outcome: Duration of Response in Portion A
Description: Duration of response: the time from first documentation of objective response (confirmed BOR of CR or PR per RECIST version 1.1) to the date of first documentation of objective progression of disease (PD) or death due to any cause. Objective PD per RECIST version 1.1: >=20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 millimeters (mm); or unequivocal progression of pre-existing lesions for non-target disease; or appearance of new lesions. This outcome measure reports the individual values for evaluable participants (instead of medians etc) due to the limited number of events.
Time Frame: as for outcome 18
Population: All participants who received at least 1 dose of PF-05082566 in Portion A and achieved an objective response. "Number analyzed" represents the number of such participants for each specified category.
Measure: Number; unit: months
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
months
  For Participant X in 0.24 mg/kg: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  For Participant X in 0.24 mg/kg |  |  |  |  |  | 5.8 |  |  |  |  |  |
  For Participant Y in 0.24 mg/kg: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  For Participant Y in 0.24 mg/kg |  |  |  |  |  | 24.2 |  |  |  |  |  |
  For Participant Z in 0.6 mg/kg: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  For Participant Z in 0.6 mg/kg |  |  |  |  |  |  |  | 22.8 |  |  |  |

20. Secondary Outcome: Time to Response in Portion A
Description: Time to response: the time from Cycle 1 Day 1 to the first documentation of objective response (confirmed BOR of CR or PR per RECIST version 1.1). BOR of CR: target lesions and non-target diseases achieved CR, without new lesions. BOR of PR: target lesions achieved CR or PR while non-target diseases were non-CR/non-PD, indeterminate or missing, and without new lesions. For target lesions, CR: complete disappearance of all target lesions except nodal disease (target nodes decreased to normal size); PR: >=30% decrease under baseline of the sum of diameters of all target measurable lesions. For non-target diseases, CR: disappearance of all non-target lesions and normalization of tumor marker levels; non-CR/non-PD: persistence of any non-target lesions and/or tumor marker level above the normal limits; Indeterminate: progression had not been determined and >=1 non-target sites were not assessed or assessment methods were inconsistent with those used at baseline.
Time Frame: as for outcome 18
Population: All participants who received at least 1 dose of PF-05082566 in Portion A and and achieved an objective response.
Measure: Median (Full Range); unit: months
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
months |  |  |  |  |  | 10.3 [2.3 to 18.4] |  | 1.8 [1.8 to 1.8] |  |  |  |

21. Secondary Outcome: Progression-Free Survival in Portion A
Description: Progression-free survival: the time from Cycle 1 Day 1 to the date of the first documentation of objective PD or death due to any cause, whichever occurred first. Objective PD per RECIST version 1.1: >=20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 mm; or unequivocal progression of pre-existing lesions for non-target disease; or appearance of new lesions.
Time Frame: as for outcome 18
Population: All participants who received at least 1 dose of PF-05082566 in Portion A and had tumor assessments.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 1 | 42 | 3 | 4 | 31 | 5 | 6 | 11
months | 1.7 [1.1 to 1.8] | 3.6 [1.7 to 5.5] | 1.7 [1.6 to 2.1] | 3.5 [1.6 to NA] — The upper limit of 95% confidence interval (CI) was not estimable due to the small number of events. | 1.7 [NA to NA] — 95% CI was not estimable due to the small number of events. | 2.1 [1.8 to 3.7] | 1.6 [1.6 to 1.6] | 3.5 [1.4 to NA] — The upper limit of 95% CI was not estimable due to the small number of events. | 1.7 [1.5 to 1.8] | 1.1 [0.2 to 1.7] | 3.3 [0.3 to NA] — The upper limit of 95% CI was not estimable due to the small number of events. | 1.8 [0.9 to 1.9]

22. Secondary Outcome: Overall Survival in Portion A
Description: Overall survival was defined as the time from Cycle 1 Day 1 to the date of death due to any cause.
Time Frame: as for outcome 18
Population: All participants who received at least 1 dose of PF-05082566 in Portion A and had tumor assessments.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 1 | 42 | 3 | 4 | 31 | 5 | 6 | 11
months | 4.6 [2.1 to 6.2] | 4.0 [3.6 to 29.7] | 7.6 [4.2 to NA] — Not estimable due to the small number of events. | 13.3 [5.9 to 24.1] | 5.9 [NA to NA] — Not estimable due to the small number of events. | 9.0 [5.8 to 16.4] | 24.5 [1.6 to NA] — Not estimable due to the small number of events. | NA [3.9 to NA] — Not estimable due to the small number of events. | 7.6 [2.9 to 12.7] | 11.2 [3.7 to NA] — Not estimable due to the small number of events. | 29.5 [1.8 to NA] — Not estimable due to the small number of events. | 6.1 [3.9 to 7.5]

23. Secondary Outcome: Number of Participants With Treatment-Emergent AEs and SAEs in Portion B
Description: as for outcome 3
Time Frame: Up to approximately 4 years
Population: All participants who received at least 1 dose of study treatment (PF-05082566 and/or rituximab) in Portion B.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 4 | 32 | 3 | 5 | 4
Participants
  AEs | 3 | 3 | 4 | 3 | 3 | 3 | 4 | 30 | 3 | 4 | 4
  SAEs | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 3 | 0 | 0 | 0
  AEs related to PF-05082566 | 2 | 2 | 2 | 2 | 1 | 2 | 3 | 17 | 2 | 1 | 1
  SAEs related to PF-05082566 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AEs related to rituximab | 3 | 2 | 3 | 3 | 2 | 2 | 3 | 17 | 2 | 3 | 3
  SAEs related to rituximab | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Number of Participants With Treatment-Emergent AEs by Maximum NCI CTCAE Grade in Portion B
Description: as for outcome 4
Time Frame: Up to approximately 4 years
Population: All participants who received at least 1 dose of study treatment (PF-05082566 and/or rituximab) in Portion B.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 4 | 32 | 3 | 5 | 4
Participants
  Grade 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 7 | 1 | 3 | 1
  Grade 2 | 0 | 2 | 2 | 0 | 0 | 2 | 2 | 17 | 1 | 1 | 3
  Grade 3 | 2 | 1 | 1 | 3 | 2 | 0 | 0 | 5 | 1 | 0 | 0
  Grade 4 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With Hematology Laboratory Abnormalities by Maximum NCI CTCAE Grade in Portion B
Description: as for outcome 5
Time Frame: Up to approximately 2 years
Population: All participants who received at least 1 dose of study treatment (PF-05082566 and/or rituximab) in Portion B and had hematology laboratory test data.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 32 | 3 | 5 | 4
Participants
  Anemia, Grade 1 | 3 | 2 | 2 | 2 | 1 | 1 | 2 | 16 | 0 | 5 | 1
  Anemia, Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 0
  Hemoglobin increased, Grade 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count increased, Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Lymphopenia, Grade 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 8 | 0 | 1 | 1
  Lymphopenia, Grade 2 | 1 | 3 | 3 | 1 | 0 | 0 | 1 | 9 | 2 | 3 | 0
  Lymphopenia, Grade 3 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 8 | 0 | 1 | 2
  Neutrophils (absolute), Grade 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0
  Neutrophils (absolute), Grade 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
  Neutrophils (absolute), Grade 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Neutrophils (absolute), Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Platelets, Grade 1 | 1 | 1 | 1 | 2 | 1 | 0 | 2 | 11 | 3 | 1 | 0
  Platelets, Grade 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Platelets, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  White blood cells, Grade 1 | 1 | 1 | 2 | 2 | 0 | 1 | 1 | 11 | 1 | 0 | 0
  White blood cells, Grade 2 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 6 | 0 | 1 | 0
  White blood cells, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0

26. Secondary Outcome: Number of Participants With Chemistries Laboratory Abnormalities by Maximum NCI CTCAE Grade in Portion B
Description: as for outcome 6
Time Frame: Up to approximately 2 years
Population: All participants who received at least 1 dose of study treatment (PF-05082566 and/or rituximab) in Portion B and had chemistries laboratory test data.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 32 | 3 | 5 | 4
Participants
  ALT, Grade 1 | 1 | 2 | 0 | 1 | 0 | 1 | 2 | 7 | 1 | 0 | 0
  ALT, Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  ALT, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Alkaline phosphatase, Grade 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 6 | 1 | 0 | 0
  AST, Grade 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 8 | 1 | 0 | 0
  AST, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Bilirubin (total), Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Bilirubin (total), Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine, Grade 1 | 2 | 3 | 4 | 2 | 3 | 3 | 2 | 27 | 3 | 4 | 4
  Creatinine, Grade 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
  Hypercalcemia, Grade 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
  Hyperglycemia, Grade 1 | 2 | 2 | 3 | 1 | 2 | 2 | 2 | 9 | 1 | 2 | 0
  Hyperglycemia, Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 0 | 1 | 1
  Hyperglycemia, Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Hyperkalemia, Grade 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 1
  Hyperkalemia, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Hyperkalemia, Grade 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia, Grade 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
  Hypermagnesemia, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypernatremia, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hypernatremia, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hypoalbuminemia, Grade 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 5 | 1 | 0 | 0
  Hypoalbuminemia, Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypocalcemia, Grade 1 | 0 | 2 | 2 | 2 | 1 | 0 | 1 | 10 | 1 | 1 | 1
  Hypocalcemia, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hypocalcemia, Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia, Grade 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0
  Hypoglycemia, Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia, Grade 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 8 | 1 | 1 | 0
  Hypomagnesemia, Grade 1 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 3 | 0 | 1 | 1
  Hyponatremia, Grade 1 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 9 | 2 | 2 | 1
  Hyponatremia, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypophosphatemia, Grade 2 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 8 | 1 | 1 | 0
  Hypophosphatemia, Grade 3 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With Clinically Significant Vital Sign Abnormalities in Portion B
Description: For vital signs in Portion B, blood pressure, pulse rate, and body temperature were measured. Clinical significance was determined by the investigator.
Time Frame: Up to approximately 2 years
Population: All participants who received at least 1 dose of study treatment (PF-05082566 and/or rituximab) in Portion B.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 4 | 32 | 3 | 5 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: PF-05082566 Cmax in Portion B
Description: Cmax of PF-05082566 was observed directly from data.
Time Frame: Cycle 1 Day 1 pre-dose, 1.5, 2, 6, 24, 48, 144, 312, and 504 hours post-dose; Cycle 2 Day 1 pre-dose, 1.5, 2, 6, 24, 48, 168, 336, and 504 hours post-dose.
Population: All participants who received at least 1 dose of PF-05082566 in Portion B and had at least 1 of the PK parameters of interest. "Number Analyzed" represents those participants who had data for each specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 30 | 3 | 5 | 4
μg/mL
  Cycle 1 | 0.6284 (11) | 1.569 (12) | 2.673 (26) | 4.167 (12) | 4.512 (29) | 7.435 (9) | 12.16 (9) | 19.20 (27) | 42.61 (26) | 89.06 (23) | 196.2 (22)
  Cycle 2: number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 27 | 3 | 5 | 4
  Cycle 2 | 0.6838 (18) | 1.948 (6) | 3.102 (18) | 3.934 (28) | 4.607 (30) | 6.481 (10) | 13.97 (24) | 20.03 (32) | 44.35 (19) | 95.16 (19) | 206.0 (29)

29. Secondary Outcome: PF-05082566 Ctrough in Portion B
Description: Ctrough of PF-05082566 was observed directly from data.
Time Frame: Day 1 pre-dose of Cycle 2
Population: All participants who received at least 1 dose of PF-05082566 in Portion B and had data for Ctrough.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 27 | 3 | 5 | 4
μg/mL | 0.1267 (47) | 0.2853 (23) | 0.3922 (29) | 0.4698 (53) | 0.3539 (110) | 0.6001 (48) | 1.486 (90) | 1.452 (62) | 5.560 (29) | 12.16 (63) | 31.34 (36)

30. Secondary Outcome: PF-05082566 Tmax in Portion B
Description: Tmax of PF-05082566 was observed directly from data as time of Cmax.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Median (Full Range); unit: hr
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 30 | 3 | 5 | 4
hr
  Cycle 1 | 1.50 [1.28 to 2.00] | 1.52 [1.00 to 1.83] | 1.06 [0.950 to 1.42] | 2.00 [1.50 to 2.00] | 1.52 [1.02 to 1.63] | 1.17 [1.00 to 1.52] | 2.00 [1.00 to 6.07] | 1.06 [0.933 to 5.45] | 2.00 [1.00 to 6.00] | 2.00 [1.50 to 6.00] | 2.00 [1.00 to 6.10]
  Cycle 2: number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 27 | 3 | 5 | 4
  Cycle 2 | 1.05 [1.00 to 1.05] | 1.08 [1.00 to 1.55] | 1.04 [1.03 to 1.08] | 1.57 [1.07 to 21.1] | 1.00 [0.967 to 1.10] | 1.50 [0.967 to 1.50] | 1.33 [1.17 to 1.50] | 1.02 [0.967 to 1.98] | 1.50 [1.50 to 1.55] | 1.50 [1.00 to 1.50] | 1.28 [1.00 to 1.50]

31. Secondary Outcome: PF-05082566 AUClast in Portion B
Description: AUClast of PF-05082566 was determined by linear/log trapezoidal method.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 30 | 3 | 5 | 4
μg*hr/mL
  Cycle 1: number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 29 | 3 | 5 | 4
  Cycle 1 | 121.1 (26) | 342.6 (13) | 513.7 (20) | 854.1 (31) | 701.7 (72) | 1130 (14) | 2373 (37) | 2772 (63) | 7955 (30) | 17120 (33) | 38180 (18)
  Cycle 2: number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 5 | 3 | 5 | 4
  Cycle 2 | 176.2 (26) | 471.5 (7) | 696.5 (17) | 1146 (35) | 733.7 (85) | 1511 (10) | 3013 (70) | 6193 (22) | 10970 (44) | 19410 (37) | 48540 (27)

32. Secondary Outcome: PF-05082566 AUCinf in Portion B
Description: as for outcome 12
Time Frame: Cycle 1 Day 1 pre-dose, 1.5, 2, 6, 24, 48, 144, 312, and 504 hours post-dose.
Population: All participants who received at least 1 dose of PF-05082566 in Portion B and had AUCinf data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 2 | 1 | 2 | 3 | 3 | 3 | 1 | 23 | 2 | 2 | 2
μg*hr/mL | 137.8 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 407.0 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 615.5 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 1076 (38) | 824.1 (78) | 1421 (24) | 2070 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 3703 (37) | 9439 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 16790 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 48870 (NA) — Geometric CV was not calculated when there were less than 3 participants with data.

33. Secondary Outcome: PF-05082566 AUCtau in Portion B
Description: AUCtau of PF-05082566 was determined using linear/log trapezoidal method.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 30 | 3 | 5 | 4
μg*hr/mL
  Cycle 1: number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 26 | 3 | 5 | 4
  Cycle 1 | 125.0 (23) | 345.0 (16) | 514.5 (21) | 871.6 (32) | 712.0 (71) | 1128 (15) | 2361 (39) | 3206 (32) | 8001 (29) | 17290 (32) | 38860 (17)
  Cycle 2: number analyzed (Participants) | 3 | 2 | 4 | 3 | 2 | 3 | 3 | 3 | 3 | 4 | 4
  Cycle 2 | 178.2 (26) | 453.9 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 701.8 (18) | 1072 (33) | 854.5 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 1521 (10) | 3116 (63) | 5967 (30) | 10220 (30) | 18150 (39) | 48030 (16)

34. Secondary Outcome: PF-05082566 CL in Portion B
Description: CL = Dose/AUCinf for Cycle 1 and Dose/AUCtau for Cycle 2.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr/kg
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 30 | 3 | 5 | 4
mL/hr/kg
  Cycle 1: number analyzed (Participants) | 2 | 1 | 2 | 3 | 3 | 3 | 1 | 23 | 2 | 2 | 2
  Cycle 1 | 0.2178 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.1470 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.1950 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.1667 (38) | 0.2911 (78) | 0.2107 (24) | 0.2900 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.3241 (37) | 0.2546 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.2973 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.2048 (NA) — Geometric CV was not calculated when there were less than 3 participants with data.
  Cycle 2: number analyzed (Participants) | 3 | 2 | 4 | 3 | 2 | 3 | 3 | 3 | 3 | 4 | 4
  Cycle 2 | 0.1683 (26) | 0.1325 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.1710 (18) | 0.1681 (33) | 0.2807 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 0.1976 (11) | 0.1928 (63) | 0.2011 (30) | 0.2351 (29) | 0.2756 (39) | 0.2080 (16)

35. Secondary Outcome: PF-05082566 Vss in Portion B
Description: Vss = CL × MRT, where CL is clearance and MRT is the mean residence time after intravenous administration.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 30 | 3 | 5 | 4
mL/kg
  Cycle 1: number analyzed (Participants) | 2 | 1 | 2 | 3 | 3 | 3 | 1 | 23 | 2 | 2 | 2
  Cycle 1 | 81.87 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 78.60 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 79.93 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 66.90 (24) | 93.68 (54) | 85.12 (4) | 126.0 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 102.8 (20) | 130.9 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 98.98 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 94.08 (NA) — Geometric CV was not calculated when there were less than 3 participants with data.
  Cycle 2: number analyzed (Participants) | 0 | 0 | 1 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2
  Cycle 2 |  |  | 81.90 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 65.42 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 85.51 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 66.27 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 100.5 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 86.99 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 94.00 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 102.2 (NA) — Geometric CV was not calculated when there were less than 3 participants with data. | 95.89 (NA) — Geometric CV was not calculated when there were less than 3 participants with data.

36. Secondary Outcome: Rituximab Cmax and Ctrough in Portion B
Description: Cmax and Ctrough of rituximab were observed directly from data.
Time Frame: Day 1 pre-dose of Cycle 2
Population: All participants who received at least 1 dose of rituximab in Portion B and had Cmax or Ctrough data for rituximab. No data were collected for this Outcome Measure.
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

37. Secondary Outcome: Number of Participants With Positive ADA for PF-05082566 and Rituximab in Portion B
Description: ADA for PF-05082566 and rituximab was detected using electrochemiluminescence assay. Positive ADA for PF-05082566: titer>=6.23. Positive ADA for rituximab: titer>=1.88.
Time Frame: Up to approximately 2 years
Population: All participants who received at least 1 dose of study treatment (PF-05082566 and/or rituximab) in Portion B and was tested for ADA. "Number Analyzed" represents those participants who had data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 4 | 32 | 3 | 5 | 4
Participants
  For PF-05082566: number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 32 | 3 | 5 | 4
  For PF-05082566 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  For rituximab | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

38. Secondary Outcome: Number of Participants With QTc Interval Meeting Categorical Summarization Criteria in Portion B
Description: Categorical summarization criteria for QTc interval: 1) absolute value of >450 to <=480 milliseconds (msec), >480 to <=500 msec, >500 msec; 2) a maximum change from baseline of >30 to <=60 msec or >60 msec.
Time Frame: Up to approximately 2 years
Population: All participants who received at least 1 dose of study treatment (PF-05082566 and/or rituximab) in Portion B and had post-baseline QTc data. "Number Analyzed" represents those participants who had data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 3 | 3 | 4 | 32 | 2 | 4 | 2
Participants
  QTc >450 to <=480 msec | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 14 | 0 | 2 | 0
  QTc >480 to <=500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  QTc >500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  QTc change >30 to <=60 msec: number analyzed (Participants) | 3 | 3 | 4 | 2 | 3 | 3 | 4 | 31 | 2 | 4 | 2
  QTc change >30 to <=60 msec | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0
  QTc change >60 msec: number analyzed (Participants) | 3 | 3 | 4 | 2 | 3 | 3 | 4 | 31 | 2 | 4 | 2
  QTc change >60 msec | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

39. Secondary Outcome: Percentage of Participants Achieving Objective Response Per Cheson 2007 Criteria in Portion B
Description: Objective Response in Portion B was defined as BOR of CR or PR according to Cheson 2007 criteria. BOR of CR or PR per Cheson 2007: CR or PR of index lesions (complete disappearance of all detectable clinical and radiographic evidence of disease, all lymph nodes returned to normal size, spleen and/or liver if enlarged prior to therapy became normal or no longer palpable; or >=50% decrease in the sum of the product diameters [SPD] of up to 6 index lesions, no increase in size of other nodes, liver or spleen), without PD of non-index lesions (ie, without: new nonnodal lesion, new nodal lesion >=15 mm in greatest transverse diameter [GTD], unequivocal progression of existing non index lesions, bone marrow that was negative and is now positive, new circulating lymphoma cells in blood cell count and/or pleural fluid, new circulating blasts in the blood cell count), and without any new lesions.
Time Frame: as for outcome 18
Population: All participants who received at least 1 dose of study treatment (PF-05082566 and/or rituximab) in Portion B and had tumor assessments for lymphoma.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 4 | 31 | 3 | 5 | 4
percentage of participants | 33.3 [0.8 to 90.6] | 0 [0 to 70.8] | 25.0 [0.6 to 80.6] | 66.7 [9.4 to 99.2] | 0 [0 to 70.8] | 0 [0 to 70.8] | 0 [0 to 60.2] | 25.8 [11.9 to 44.6] | 33.3 [0.8 to 90.6] | 20.0 [0.5 to 71.6] | 0 [0 to 60.2]

40. Secondary Outcome: Duration of Response in Portion B
Description: Duration of Response in Portion B was defined, for participants with an objective response (BOR of CR or PR per Cheson 2007 criteria), as the time from first documentation of objective response to the date of first documentation of objective PD or death due to any cause. Objective PD per Cheson 2007 was defined as: PD of index lesions (>=50% increase in SPD of previously involved sites from nadir), or PD of non-index lesions (new nonnodal lesion, new nodal lesion >=15 mm in GTD, unequivocal progression of existing non index lesions, bone marrow that was negative and is now positive, new circulating lymphoma cells in blood cell count and/or pleural fluid, new circulating blasts in the blood cell count), or appearance of new lesions.
Time Frame: as for outcome 18
Population: All participants who received at least 1 dose of study treatment (PF-05082566 and/or rituximab) in Portion B, had tumor assessments for lymphoma, and achieved an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 8 | 1 | 1 | 0
months | NA [NA to NA] — The median estimates of time to event, upper and lower limits of 95% CI were not estimable due to the small number of events. |  | NA [NA to NA] — The median estimates of time to event, upper and lower limits of 95% CI were not estimable due to the small number of events. | NA [8.0 to NA] — The median estimates of time to event and upper limit of 95% CI were not estimable due to the small number of events. |  |  |  | 12.0 [2.1 to NA] — Not estimable due to the small number of events. | 9.5 [NA to NA] — Not estimable due to the small number of events. | NA [NA to NA] — The median estimates of time to event, upper and lower limits of 95% CI were not estimable due to the small number of events. |

41. Secondary Outcome: Time to Response in Portion B
Description: Time to response in Portion B was defined, for participants with an objective response (BOR of CR or PR per Cheson 2007 criteria), as the time from Cycle 1 Day 1 to the first documentation of objective response. BOR of CR or PR per Cheson 2007: CR or PR of index lesions (complete disappearance of all detectable clinical and radiographic evidence of disease, all lymph nodes returned to normal size, spleen and/or liver if enlarged prior to therapy became normal or no longer palpable; or >=50% decrease in the SPD of up to 6 index lesions, no increase in size of other nodes, liver or spleen), without PD of non-index lesions (ie, without: new nonnodal lesion, new nodal lesion >=15 mm in GTD, unequivocal progression of existing non index lesions, bone marrow that was negative and is now positive, new circulating lymphoma cells in blood cell count and/or pleural fluid, new circulating blasts in the blood cell count), and without any new lesions.
Time Frame: as for outcome 18
Population: as for outcome 40
Measure: Median (Full Range); unit: months
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 8 | 1 | 1 | 0
months | 2.1 [2.1 to 2.1] |  | 2.1 [2.1 to 2.1] | 2.0 [1.9 to 2.1] |  |  |  | 2.1 [1.9 to 2.2] | 3.9 [3.9 to 3.9] | 7.4 [7.4 to 7.4] |

42. Secondary Outcome: Progression-Free Survival in Portion B
Description: Progression-free survival in Portion B was defined as the time from Cycle 1 Day 1 to the date of the first documentation of objective PD (per Cheson 2007) or death due to any cause, whichever occurred first. Objective PD per Cheson 2007 was defined as: PD of index lesions (>=50% increase in SPD of previously involved sites from nadir), or PD of non-index lesions (new nonnodal lesion, new nodal lesion >=15 mm in GTD, unequivocal progression of existing non index lesions, bone marrow that was negative and is now positive, new circulating lymphoma cells in blood cell count and/or pleural fluid, new circulating blasts in the blood cell count), or appearance of new lesions.
Time Frame: as for outcome 18
Population: as for outcome 39
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 4 | 31 | 3 | 5 | 4
months | NA [7.4 to NA] — The median estimates of time to event and upper limit of 95% CI were not estimable due to the small number of events. | 8.1 [1.9 to 8.1] | 11.8 [3.9 to NA] — The upper limit of 95% CI was not estimable due to the small number of events. | 9.9 [6.0 to NA] — The upper limit of 95% CI was not estimable due to the small number of events. | 2.1 [1.8 to 2.1] | 5.7 [3.9 to NA] — The upper limit of 95% CI was not estimable due to the small number of events. | 4.8 [0.7 to 9.4] | 3.9 [2.1 to 5.7] | 16.3 [13.4 to 19.2] | 3.9 [2.1 to NA] — The upper limit of 95% CI was not estimable due to the small number of events. | 3.0 [2.1 to 4.2]

43. Secondary Outcome: Overall Survival in Portion B
Description: Overall survival was defined as the time from Cycle 1 Day 1 to the date of death due to any cause.
Time Frame: as for outcome 18
Population: as for outcome 39
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 3 | 4 | 31 | 3 | 5 | 4
months | NA [NA to NA] — Not estimable due to the small number of events. | NA [NA to NA] — Not estimable due to the small number of events. | NA [NA to NA] — Not estimable due to the small number of events. | NA [NA to NA] — Not estimable due to the small number of events. | NA [9.6 to NA] — Not estimable due to the small number of events. | 50.2 [NA to NA] — Not estimable due to the small number of events. | NA [0.7 to NA] — Not estimable due to the small number of events. | NA [18.0 to NA] — Not estimable due to the small number of events. | NA [39.5 to NA] — Not estimable due to the small number of events. | NA [5.4 to NA] — Not estimable due to the small number of events. | NA [4.9 to NA] — Not estimable due to the small number of events.

44. Other Pre Specified Outcome: Biomarkers Linked With Immunomodulation and Cytokine Release
Description: This was an exploratory endpoint and no data were collected.
Time Frame: Days 1, 14, 29 and 57
Population: This was an exploratory endpoint and no data were collected.
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

45. Other Pre Specified Outcome: Exploratory Pharmacodynamic Biomarkers
Description: This was an exploratory endpoint and no data were collected.
Time Frame: Days 1 and 21
Population: This was an exploratory endpoint and no data were collected.
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

46. Other Pre Specified Outcome: Patient-Reported Outcomes of PF-05082566 and Rituximab When Given in Combination in Follicular Lymphoma Participants
Description: This was an exploratory endpoint and was not evaluated. Patient-reported outcome questionnaires were not completed as a result of administrative processing error.
Time Frame: Up to 2 years
Population: This was an exploratory endpoint and was not evaluated. Patient-reported outcome questionnaires were not completed as a result of administrative processing error.
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 4 years.
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Portion A: PF-05082566 0.006mg/kg | Portion A: PF-05082566 0.03mg/kg | Portion A: PF-05082566 0.06mg/kg | Portion A: PF-05082566 0.12mg/kg | Portion A: PF-05082566 0.18mg/kg | Portion A: PF-05082566 0.24mg/kg | Portion A: PF-05082566 0.3mg/kg | Portion A: PF-05082566 0.6mg/kg | Portion A: PF-05082566 1.2mg/kg | Portion A: PF-05082566 2.4mg/kg | Portion A: PF-05082566 5mg/kg | Portion A: PF-05082566 10mg/kg | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2
All-Cause Mortality (participants affected / at risk) | 4/4 | 3/3 | 5/6 | 3/4 | 1/3 | 27/42 | 2/3 | 2/4 | 21/31 | 2/5 | 3/6 | 9/11 | 0/3 | 0/3 | 0/4 | 0/3 | 1/3 | 1/3 | 2/4 | 8/32 | 1/3 | 2/5 | 2/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 2/6 | 1/4 | 0/3 | 13/42 | 0/3 | 0/4 | 8/31 | 1/5 | 2/6 | 3/11 | 1/3 | 0/3 | 0/4 | 2/3 | 1/3 | 1/3 | 1/4 | 3/32 | 0/3 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 3/3 | 5/6 | 4/4 | 3/3 | 36/42 | 3/3 | 4/4 | 23/31 | 4/5 | 5/6 | 9/11 | 3/3 | 3/3 | 4/4 | 3/3 | 3/3 | 3/3 | 3/4 | 29/32 | 3/3 | 4/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Portion A: PF-05082566 0.006mg/kg (N=4) | Portion A: PF-05082566 0.03mg/kg (N=3) | Portion A: PF-05082566 0.06mg/kg (N=6) | Portion A: PF-05082566 0.12mg/kg (N=4) | Portion A: PF-05082566 0.18mg/kg (N=3) | Portion A: PF-05082566 0.24mg/kg (N=42) | Portion A: PF-05082566 0.3mg/kg (N=3) | Portion A: PF-05082566 0.6mg/kg (N=4) | Portion A: PF-05082566 1.2mg/kg (N=31) | Portion A: PF-05082566 2.4mg/kg (N=5) | Portion A: PF-05082566 5mg/kg (N=6) | Portion A: PF-05082566 10mg/kg (N=11) | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 (N=3) | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 (N=3) | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 (N=4) | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 (N=3) | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 (N=3) | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 (N=3) | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 (N=4) | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 (N=32) | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 (N=3) | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 (N=5) | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2 (N=4)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Portion A: PF-05082566 0.006mg/kg (N=4) | Portion A: PF-05082566 0.03mg/kg (N=3) | Portion A: PF-05082566 0.06mg/kg (N=6) | Portion A: PF-05082566 0.12mg/kg (N=4) | Portion A: PF-05082566 0.18mg/kg (N=3) | Portion A: PF-05082566 0.24mg/kg (N=42) | Portion A: PF-05082566 0.3mg/kg (N=3) | Portion A: PF-05082566 0.6mg/kg (N=4) | Portion A: PF-05082566 1.2mg/kg (N=31) | Portion A: PF-05082566 2.4mg/kg (N=5) | Portion A: PF-05082566 5mg/kg (N=6) | Portion A: PF-05082566 10mg/kg (N=11) | Portion B: PF-05082566 0.03mg/kg + Rituximab 375mg/m^2 (N=3) | Portion B: PF-05082566 0.06mg/kg + Rituximab 375mg/m^2 (N=3) | Portion B: PF-05082566 0.12mg/kg + Rituximab 375mg/m^2 (N=4) | Portion B: PF-05082566 0.18mg/kg + Rituximab 375mg/m^2 (N=3) | Portion B: PF-05082566 0.24mg/kg + Rituximab 375mg/m^2 (N=3) | Portion B: PF-05082566 0.3mg/kg + Rituximab 375mg/m^2 (N=3) | Portion B: PF-05082566 0.6mg/kg + Rituximab 375mg/m^2 (N=4) | Portion B: PF-05082566 1.2mg/kg + Rituximab 375mg/m^2 (N=32) | Portion B: PF-05082566 2.4mg/kg + Rituximab 375mg/m^2 (N=3) | Portion B: PF-05082566 5mg/kg + Rituximab 375mg/m^2 (N=5) | Portion B: PF-05082566 10mg/kg + Rituximab 375mg/m^2 (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 5 (7) | 1 (1) | 1 (1) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 6 (8) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (8) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 9 (10) | 0 (0) | 0 (0) | 10 (11) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 1 (1) | 1 (2) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 18 (19) | 0 (0) | 2 (2) | 8 (10) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 6 (7) | 0 (0) | 2 (3) | 1 (1)
Implant site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 9 (11) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 6 (7) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 1 (1) | 1 (3) | 3 (3) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (5) | 0 (0) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 7 (7) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 8 (10) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT01307267/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT01307267/SAP_001.pdf